CLINICAL TRIAL: NCT05514093
Title: Beyond Silence: Advancing E-mental Health Solutions to Support Canadian Healthcare Workers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14740
Record Dates: First submitted 2022-08-09; First posted 2022-08-24 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Issue; Mental Stress; Post-traumatic Stress Disorder; Moral Injury
Keywords: Mental health; Peer support; Mobile health; Healthcare workers
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- App users: As this is a single cohort study, there is only one group consisting of the Beyond Silence app users.
  Interventions: Device: Beyond Silence App

INTERVENTIONS:
Device: Beyond Silence App — The Beyond Silence app is designed to be a "mental health coach in your pocket" for healthcare workers. It provides opportunities to build mental health literacy and reduce barriers to seeking support, including access to peer support either within or outside the organization.
  Other Names: Beyond Silence

SUMMARY:
The purpose of this project is to scale implementation and evaluation of an m-health app designed to promote early intervention and mental health support for frontline healthcare workers to reduce their risk of post-traumatic stress disorder (PTSD) and/or the mental health impact of the COVID-19 pandemic. Beyond Silence has received an additional year of funding to scale implementation across 4-6 additional healthcare organizations.

DETAILED DESCRIPTION:
This project was designed to respond to the urgent and critical need for accessible mental health services and supports for front-line healthcare workers. Innovative solutions are needed to ensure the psychological health and safety of frontline workers and to ensure quality care for the millions of Canadians who relied on their services. This project provides an opportunity to study the implementation and impact of Beyond Silence, a new e-mental health approach to early intervention and peer support that was customized for healthcare workers.

The objectives of this study are to answer both implementation and impact questions:

Implementation:

1. What are the patterns of app use among healthcare workers over a 3-6 month period?
2. What factors influence how the app is utilized among workers in diverse healthcare organizations?

   Impact:
3. Does use of the app increase mental health literacy among healthcare workers?
4. Does the app increase outreach to peer support?
5. Does outreach to peer support in the app reduce the level of distress?

This is a prospective cohort implementation study, studying the implementation and impact of the app over a 3-6 month period in participating healthcare organizations. The Consolidated Framework for Implementation Research (CFIR) informs the exploration of how the app is adopted and the individual and organizational forces that shape adoption. Pre/post impact data are being collected over the implementation period to assess whether the app leads to improved mental health knowledge among workers who use the app (primary outcome), and to increased access to peer support (secondary outcome).

Recruitment for this study is occuring on three levels: (1) organization (2) peer support providers (3) frontline healthcare workers. Eight to ten healthcare organizations across Canada have been recruited into the study, with at least one organizational champion who liaises with the research team. Champions are interviewed to understand the workplace context and create a communication plan. Each organization also nominates at least 4-5 peer support providers who are trained to provide service through the app. Frontline workers are invited to complete a baseline survey, then invited to download the app using an organizational code. Implementation takes place over a 3-6 month period; utilization patterns are tracked over time (aggregate data only). At the end of the trial, champions will be interviewed again to gather their feedback, and peer support providers will be invited to a focus group discussion to reflect on the implementation process. All employees are invited to complete a follow-up survey to gather their input and to track changes in mental health knowledge, mental distress, and help outreach. Implementation and impact data will be analyzed to identify trends within and across organizations.

The investigators are utilizing a multi-pronged approach to data collection via the following:

1. App utilization data including adoption rates across each organization, as well as aggregate data on how often the app was used, average duration of use, the number of times different features were accessed, and how often users accessed links to the different types of peer support.
2. App user impact - impact on app users is tracked through baseline and follow-up surveys to see if there are any statistically significant changes in mental health literacy, symptoms of mental distress (anxiety, depression, PTSD), burn-out, help outreach behaviours, and perceived psychological safety.
3. Peer support provider focus group interviews will be conducted after the implementation period to explore providers' experiences facilitating peer support via the app.
4. Organizational champion interviews will be conducted after the implementation period to explore organizational contextual factors.

Analysis of the collected survey data will examine change scores across the dataset as well as trends, with results disaggregated by gender, caregiver status, work role, organization, job tenure. Linear mixed models will be used to track changes over time in mental health knowledge (primary outcome), distress levels, and self-report of help-seeking/outreach. The model includes a fixed effect for time and random effects for organization types and participants. Age, gender, and caregiver status will be included in the models as covariates. The investigators also will explore potential predictors of outcomes using linear regression models (e.g., app usage, age, gender, education, role in organization - clinical/non-clinical). Additionally, qualitative content analysis will be used to examine focus group and interview data. All focus group and interview data are transcribed with the transcripts then reviewed and used for thematic analysis. Lastly, a cost-benefit analysis will be conducted to examine app implementation costs.

ELIGIBILITY:
Inclusion Criteria:

* Employees (full-time or part-time) at participating healthcare organizations
* Agree to download the Beyond Silence app to their mobile phone (Apple or Android)

Exclusion Criteria:

* Not able to access app on their smart device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthcare workers of all ages and genders (from frontline workers to middle and high-level management) in the participating organizations. Frontline healthcare workers include any staff providing direct patient services (e.g., personal support workers, healthcare aids, nursing. physician, allied health) as well as non-clinical staff (e.g. management, administration).
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline mental health literacy after implementation | Baseline, 3-6 months
  The primary outcome is changes in mental health knowledge scores from baseline to follow-up among app users. Mental health literacy regarding how to identify and address mental health issues in the workplace will be rated on a 7-point scale of perceived knowledge.

SECONDARY OUTCOMES:
Change from baseline depression after implementation | Baseline, 3-6 months
  Depression will be assessed via the Patient Health Questionnaire-2 (PHQ-2), a brief and valid two item screening tool for the core symptoms depression
Change from baseline anxiety after implementation | Baseline, 3-6 months
  Symptoms of anxiety will be measured using the Generalized Anxiety Disorder Assessment-7 (GAD-7), which consists of seven questions answered via a 4-point Likert scale
Change from baseline post-traumatic stress disorder after implementation | Baseline, 3-6 months
  To assess PTSD, the PTSD Checklist for Diagnostic and Statistics Manual 5 (PCL-5) will be used, a 20-item standardized self-report measure that assesses the DSM-5 symptoms of PTSD over the past month
Change from baseline burn-out after implementation | Baseline, 3-6 months
  To assess mental distress related to burnout, the Maslach Burnout Inventory-2 (MBI-2) will be used. This validated burn-out screening tool consists of two questions answered via a 7-point Likert scale.
Change from baseline perceived psychological health and safety after implementation | Baseline, 3-6 months
  Perceived psychological health and safety in the workplace will be assessed via excerpts from StressAssess, a tool based on the Copenhagen validated Canadian survey. We are utilizing 13 questions from this survey, which are answered via variable Likert scale responses.
Change from baseline help outreach behavior after implementation | Baseline, 3-6 months
  Participants will be asked whether they have sought help for themselves or a colleague in the past 3 months. If yes, they will be asked to identify the type of help sought.
Peer support | 3-to-6-month implementation period
  Following use of peer support services, app users will be invited to fill out an in-app survey immediately following the peer support interaction, asking service recipients to rate how they felt before and after the interaction (10-point Likert scale) and to comment on their experience.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada